CLINICAL TRIAL: NCT05322265
Title: Complication in Laparoscopic Renal and Adrenal Surgery (CLARAS): an International Multicenter Study
Brief Title: Complication in Laparoscopic Renal and Adrenal Surgery (CLARAS)
Acronym: CLARAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Palermo (Other)
Collaborators: Fundacio Puigvert (Other)
Responsible Party: Principal Investigator, Prof. Antonino Agrusa, full professor of surgery, University of Palermo
Other Study IDs: CLARAS study
Record Dates: First submitted 2022-04-03; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Adrenal Disease; Renal Cancer; Surgery--Complications
Keywords: laparoscopic surgery; renal surgery; adrenalectomy; complication in laparoscopic surgery
MeSH Terms: conditions — Adrenal Gland Diseases; Kidney Neoplasms | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- complicated patients: patients underwent to laparoscopic renal and adrenal surgery with intraoperative complications
  Interventions: Procedure: laparoscopic surgery for renal and adrenal diseases
- uncomplicated patients: patients underwent to laparoscopic renal and adrenal surgery with no complication during surgical procedure

INTERVENTIONS:
Procedure: laparoscopic surgery for renal and adrenal diseases — type of treatment for patients underwent to laparoscopic surgery for renal and adrenal diseases with intraoperative complications
  Groups: complicated patients

SUMMARY:
the aim of this study is clarify complication and their resolution in laparoscopic renal and adrenal surgery.

DETAILED DESCRIPTION:
the aim of this study is clarify complication and their resolution in laparoscopic renal and adrenal surgery.

ELIGIBILITY:
Inclusion Criteria:

renal diseases with indication to surgery adrenal masses

Exclusion Criteria:

open surgery in principle

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients underwent to laparoscopic renal and adrenal surgery form april 2017 to march 2022 in several high volume surgical center
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
intraoperative complications | 5 years
  evaluation of intraoperative complication and their resolution

CONTACTS AND LOCATIONS:
Overall Officials: Antonino Agrusa, Medicine, Study Director — University of Palermo
Locations (1):
- University of Palermo, Palermo, Italy

IPD SHARING:
Plan to Share IPD: No